CLINICAL TRIAL: NCT06921252
Title: Does Recurrent Pancreatic Cancer Really Have Similar Outcome Compared With Primary Metastatic Pancreatic Cancer?
Status: Completed | Type: Observational
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Head of Surgery, Kochi University
Other Study IDs: Kochi University
Record Dates: First submitted 2025-03-13; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- chemotherapy for metastatic pancreatic cancer: chemotherapy
  Interventions: Drug: chemotherapy agents
- chemotherapy for recurrent pancreatic cancer: postoperative chemotherapy
  Interventions: Drug: chemotherapy agents

INTERVENTIONS:
Drug: chemotherapy agents — Overall, data of 276 patients (144 men and 132 women, 224 Rec-PC and 51 PM-PC) were retrospectively analyzed. The median patient age was 70 (range; 29-91) years. Serum carbohydrate antigen (CA) 19-9 among Rec-PC group (median; 207 U/mL) and PM-PC group (median; 1680 U/mL) was statistically different. Rec-PC patients received gemcitabine plus nab-paclitaxel (106), S-1 (37), gemcitabine (22), FOLRIFINOX (18) and other (8) regimen as a first line chemotherapy. 67 Rec-PC patients underwent any local treatment. PM-PC patients received gemcitabine plus nab-paclitaxel (34), FOLRIFINOX (8), gemcitabine (5), S-1 (2) and other (2) regimen as a first line chemotherapy.

SUMMARY:
The recurrent pancreatic cancer (Rec-PC) after radical surgery is sometimes eligible to clinical trial of chemotherapy for unresectable pancreatic cancer. However, the difference between Rec-PC and primary metastatic pancreatic cancer (PM-PC) did not know well. Thus, whether Rec-PC and PM-PC should be included in the same category when conducting clinical trials evaluating chemotherapy remains controversial. The purpose of this study is to investigate the difference of overall survival (OS) between Rec-PC and PM-PC, and analyze their impact on prognosis.

ELIGIBILITY:
Inclusion Criteria:

* unresectable pancreatic cancer

Exclusion Criteria:

* Patients expected to survive for less than three months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective database review of patients with recurrent or primary metastatic pancreatic cancer at a single institution, from 2010 to 2023, was conducted.
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of evaluation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

IPD SHARING:
Plan to Share IPD: No